CLINICAL TRIAL: NCT02018133
Title: Identification of Markers for Determining the Efficacy of Vitamin D Receptor Activator Therapy in Stage 3/4 CKD Patients
Status: Completed | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Alan Lau, Professor, University of Illinois at Chicago
Other Study IDs: 2008-0929; BMK-001 (Other: Abbott Laboratories)
Record Dates: First submitted 2012-06-20; First posted 2013-12-23 (Estimated); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: CKD Stage 3/4
Keywords: CKD; chronic; kidney; vitamin D
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Vitamin D; paricalcitol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vitamin D or Placebo: Take vitamin D for 2 weeks. 2mg daily before meal
  Interventions: Drug: Vitamin D 2mg daily for 2 weeks oral paricalcitol; Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D 2mg daily for 2 weeks oral paricalcitol — vitamin D 2 capsules daily
  Other Names: Zemplar
Drug: Placebo — placebo 2 capsule daily

SUMMARY:
The purpose of this study is to identify genes that are responsive to paricalcitol (active vitamin D) therapy. Scientists have found that over 30 different types of cells in the body respond to vitamin D therapy, including blood vessels. Low levels of vitamin D may reduce the amount of calcium in the blood, increase the amount of parathyroid hormone (PTH) and cause the parathyroid gland (small gland located in the neck) to get bigger which is called secondary hyperparathyroidism (SHPT). Also, low levels of vitamin D may worsen the heart disease seen in dialysis patients. Paricalcitol, a man-made active vitamin D, is a replacement for vitamin D for preventing and treating SHPT. Studies that followed patients on dialysis have found: (1) differences in death rates between those who received active vitamin D compared with no activated vitamin D, and (2) a survival benefit in chronic kidney disease (CKD) patients receiving paricalcitol, over calcitriol (natural active vitamin D). Researchers have considered that giving paricalcitol to people with (CKD) may also prevent or slow the progression of heart disease.

Currently, physicians can only tell how well the vitamin D is working by measuring PTH concentrations. This study aims to identify markers in the blood that can be used to determine the efficacy of Vitamin D therapy.

DETAILED DESCRIPTION:
After baseline information and laboratory tests are obtained, subjects will be randomized to receive either oral paricalcitol at 2 mcg daily for 2 weeks or placebo. After a washout period of 4 weeks, those subjects who received paricalcitol will receive placebo for 2 weeks and those who received placebo will receive paricalcitol for 2 weeks. A simple blood draw will be obtained from the patient on days 0, 1, and 14 of each treatment arm, and they will also be assessed for side effects at the end of each treatment.

The blood obtained during these visits will be analyzed for any changes that may have occurred in the white blood cells (WBC) and/or plasma. These samples will be tested to see if there are any markers in the blood that changed after treatment with vitamin D. The samples collected will be temporarily stored in the research laboratory and subsequently sent to a separate laboratory (Genus Systems Company) in batches for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease stage 3/4
* PTH: >70 pg/ml
* If on ACEI/ARB, optimized and stable dose

Exclusion Criteria:

* Failure to provide informed consent
* Prior active vitamin D oral or parenteral treatment, including calcitriol, paricalcitol and doxercalciferol
* Glomerulonephritis requiring active treatment with immunosuppressive therapy
* Serum phosphorus: > 5.2 mg/dL
* Serum calcium (corrected for albumin): > 10.0 mg/dL
* Clinical unstable medical conditions (other than CKD)
* Use of any investigational drug within the past 30 days or 5 half-lives, whichever is longer
* History of malignancy, other than basal cell carcinoma of the skin
* History of hypersensitivity to vitamin D or its analogs
* Pregnant or nursing (lactating) women
* Women of child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic kidney disease stage 3/4, with PTH >70 pg/ml and if on ACEI/ARB, the dose is optimized or stable
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2009-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
examine the gene expression pattern in white blood cells obtained from Stage 3/4 CKD patients before and after paricalcitol treatment | 2 weeks
  determine gene expression

CONTACTS AND LOCATIONS:
Overall Officials: Alan Lau, PharmD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States